CLINICAL TRIAL: NCT01411072
Title: Biomarker Directed Adjuvant Chemotherapy for Resected Pancreas Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Panc002/ethics 25823
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Pancreas Cancer
Keywords: Biomarker directed adjuvant chemotherapy; resected pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine (Experimental)
  Interventions: Drug: gemcitabine
- 5-fluorouracil (Experimental)
  Interventions: Drug: 5-fluorouracil

INTERVENTIONS:
Drug: gemcitabine — Gem 1000 mg/m2 IV weekly for 3 weeks then one week off of each 28 day cycle
  Other Names: hENT1 high group
  Arms: Gemcitabine
Drug: 5-fluorouracil — 5-FU 425 mg/m2 and Leucovorin 20 mg/m2 IV day 1, 2, 3, 4, and 5 of each 28 day cycle
  Other Names: hENT1 low group
  Arms: 5-fluorouracil

SUMMARY:
Chemotherapy is given after curative surgery for pancreas cancer to try to improve cure rates. There are two choices of chemotherapy which are currently considered equal treatments: gemcitabine or 5-fluorouracil (5FU). This study is trying to determine if one of two standard chemotherapies is better than the other depending on whether patients have high or low human equilibrative nucleoside transporter 1 (hENT1). hENT1 is a protein that is found in varying amounts on pancreas cancers.

DETAILED DESCRIPTION:
The rationale for this pilot study is based on trying to better deliver adjuvant chemotherapy by selecting treatment for patients that is individualized based on the hENT1 biomarker. Gemcitabine (gem) requires human equilibrative nucleoside transporter 1 (hENT1) to enter cells. If a pancreatic cancer has low hENT1, gem will not be able to enter cells efficiently. 5-fluorouracil (5FU) does not require the same transport into cells. Thus, upfront hENT1 testing will allow determination of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented pancreatic adenocarcinoma not previously treated with systemic therapy.
* Complete macroscopic and microscopic (R0) resection for ductal adenocarcinoma of the pancreas with no evidence of malignant ascites, peritoneal metastases or distant metastases. Lack of recurrent and/metastatic disease must be confirmed radiologically with CT chest, abdomen, and pelvis prior to enrolment.
* Adequate tissue available for IHC testing of hENT1. Histological/cytological confirmation of tissue to ensure sufficient material is available for hENT1 analysis by the Cross Cancer Institute (CCI) is required. Paraffin block sufficient for preparing ≥ 6 unstained slides for central storage and testing if required by oncologist.
* ECOG performance status of 0 - 2. (Appendix B)
* Age ≥ 18 years
* Life expectancy of at least 6 months based on discretion of treating
* Adequate hematologic function defined by the following laboratory parameters: Hemoglobin > 100, Platelet count > 100 and Absolute granulocyte count > 1.5.
* Adequate hepatic and renal function defined by the following laboratory parameters: AST and ALT ≤ 2.5 X upper limit of institutional normal, bilirubin ≤ upper limit of institutional normal, and calculated creatinine clearance of ≥ 50 mL/min using the Cockcroft-Gault formula, if just below 50 mL/min based on this formula then GFR ≥ 50 mL/min as determined.
* Patients may have received prior curative radiotherapy for a different malignancy (unless radiation was curative therapy to ≥ 25% of bone marrow stores) and patients must have recovered from the toxic effects of this treatment.
* Patients must be started on protocol ≤ 10 weeks from the date of curative surgical resection, and patients must have recovered from the toxic effects of surgery.
* Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.

Exclusion Criteria:

* Patients who have received prior chemotherapy or radiation delivered as parts of initial curative therapy for pancreas cancer (i.e. neoadjuvant or adjuvant chemotherapy administered alone and/or concurrently delivered with radiation and/or surgery) are not permitted. Metastatic patients are not permitted.
* Prior treatment for a different malignancy with > 6 cycles of traditional alkylating agent-based chemotherapy, > 2 cycles of carboplatin-based chemotherapy, or concurrent treatment with other experimental drugs or anti-cancer therapy.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, short gut syndrome, or history of bowel obstruction due to peritoneal metastases.
* Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or non-melanoma skin cancer, unless at least 5 years have elapsed since last treatment and the patient is considered cured.
* Any serious medical condition within 6 months prior to study entry such as myocardial infarction, uncontrolled congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, cerebrovascular diseases, uncontrolled hypertension, uncontrolled diabetes, uncontrolled psychiatric disorder, serious infection, active peptic ulcer disease, or other medical condition that.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Pregnant or lactating women; women of child bearing potential must have a negative serum pregnancy test within 7 days of trial registration. Women or men of child bearing potential must use effective contraception (defined by the treating physician) which must be documented in study CRFs.
* Any other reason the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Post treatment, patients will be followed every 3 months via phone call and/or electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Spratlin, MD, FRCPC, Principal Investigator — Cross Cancer Institute; Jennifer Spratlin, MD, FRCPC, Study Chair — Cross Cancer Institute
Locations (2):
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta